CLINICAL TRIAL: NCT00417911
Title: Clinical Protocol Bortezomib Consolidation in Patients With Myeloma Following Treatment With High-dose Melphalan and Autologous Stem Cell Support. A Randomised NMSG Trial (15/05)
Brief Title: Efficacy of Bortezomib Consolidation After High-dose Melphalan With Stem Cell Support in Myeloma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Myeloma Study Group (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Ulf-Henrik Melqvist, Nordic Myeloma Study Group, Sahlgrenska University Hospital Gothenborg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMSG 15/05; EudraCT No: 2005-002756-18
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; autologous stem cell transplantation; high-dose melphalan; bortezomib; consolidation; event free survival; phase III
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

ARMS (2):
- No treatment (Active Comparator)
  Interventions: Drug: bortezomib
- Bortezomib consolidation (Experimental): Bortezomib consolidation : 20 injections starting 3 months after ASCT
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Bortezomib 1,3 mg/sqm Days 1,4,8,11 for two 3-week cycles and then once a week for three weeks in 4 4-week cycles

SUMMARY:
Multiple myeloma is a malignant incurable hematological disease where survival has been significantly improved by high-dose melphalan with autologous stem cell support (ASCT) in younger patients. However, the disease will eventually relapse and new treatment is demanded. Bortezomib is a newly approved drug for treating relapsing multiple myeloma. It has a different biological effect and response even in patients refractory to conventional chemotherapy. The purpose of the study is in a randomized design to investigate if addition of bortezomib by 20 injections during a 4 months period starting 3 month after ASCT can prolong the time to progression compared to patients receiving no consolidation or maintenance therapy.

DETAILED DESCRIPTION:
Rationale:

ASCT prolongs EFS and OS for myeloma patients < 65 years of age. During the period from ASCT to progression most myeloma patients experience few symptoms and have a good quality of life11. A further prolongation of EFS would be a big step forward in myeloma treatment. Bortezomib is a new promising agent, which has shown clear anti-myeloma effect in heavily pre-treated patients. After ASCT the tumour cell burden is low and it is the hypothesis of this clinical trial that the unique mechanism of action of bortezomib may reduce the number of tumour cells even further and by doing so prolong EFS.

Primary objective:

* Evaluate the effect on EFS (an event is defined as either progression or death of any cause without preceding progression) of consolidation treatment with bortezomib after ASCT compared to no consolidation

Secondary objectives:

* Overall survival from ASCT
* Overall survival from start of relapse treatment
* Time to need for relapse treatment
* Response rate in patients not in CR following ASCT
* Toxicity from consolidation treatment
* Quality of life
* Cost utility
* Planned subgroup analysis: comparison of primary and secondary endpoint in patients receiving one vs. two high dose treatments

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic myeloma diagnosis according to criteria in attachment 3
* ASCT is performed or has been performed in the last five weeks (time limit two weeks for patients randomised at 2nd transplantation) as a part of primary therapy
* Signed informed consent given prior to any study related activities have been performed

Exclusion Criteria:

* Prior exposure to bortezomib
* Allogeneic transplantation scheduled as a part of the primary treatment
* Neuropathy > Grade 2 (neurological symptoms interfering with ADL)
* Non-secreting myeloma
* Other concurrent disease making bortezomib treatment unsuitable
* Positive pregnancy test (only applicable for women with childbearing potential)
* Has known or suspected hypersensitivity or intolerance to boron, mannitol, or heparin, if an indwelling catheter is used
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrolment, New York Heart Association (NYHA) Class III or IV heart failure (Attachment 6, NYHA Classification of Cardiac Disease), uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
* History of hypotension or has decreased blood pressure (sitting systolic blood pressure [SBP] £100 mmHg and/or sitting diastolic blood pressure [DBP] £60 mmHg)
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Have received an experimental drug or used an experimental medical device within 4 weeks prior to inclusion into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect on EFS (an event is defined as either progression or death of any cause without preceding progression) of consolidation treatment with bortezomib after ASCT compared to no consolidation | 1 year after randomization of the last patient

SECONDARY OUTCOMES:
Overall survival from ASCT
Overall survival from start of relapse treatment
Time to need for relapse treatment
Response rate in patients not in CR following ASCT
Toxicity from consolidation treatment
Quality of life
Cost utility
Planned subgroup analysis: comparison of primary and secondary endpoint in patients receiving one vs. two high dose treatments

CONTACTS AND LOCATIONS:
Overall Officials: Ulf-Henrik Mellqvist, Dr., PhD, Principal Investigator — NMSG
Locations (20):
- Denmark (5):
  - Hæmatologisk afdeling B, Aalborg Sygehus Syd, Aalborg
  - Hæmatologisk afd. B, Århus Universitetshospital, Amtssygehuset, Århus C
  - Hæmatologisk afdeling L Amtssygehuset i Herlev, Herlev
  - Medicinsk Hæmatologisk afd L4042, Rigshospitalet, København Ø
  - Hæmatologisk afd X, Odense Universitetshospital, Odense C
- Finland (2):
  - Tampere University Hospital, Dep 10a, Tampere
  - Turku University Hospital, Dept. of Medicine, PL 52,, Turku
- Hemathology department, University State Hospital, Landspitali, Reykjavik, Iceland
- Norway (5):
  - Hematologisk seksjon, med avd, Haukeland Universitetssykehus, Bergen
  - Seksjon for blodsykdommer, Med. avd.,Rikshospitalet, Oslo
  - Hematologisk avdeling Ullevål Sykehus, Oslo
  - Med avd B, Hematologisk seksjon, Universitetssykehuset Nord Norge, Tromsø
  - Hematologisk seksjon Regionssykehuset, Trondheim
- Sweden (7):
  - Hematologiska klin, Huddinge sjukhus, Huddinge
  - Hematologkliniken, Universitetssjukhuset, Linköping
  - University Hospital Lund, Lund
  - Medicinklin, Universitetssjukhuset MAS,, Malmo
  - Medicinkliniken, Universitetssjukhuset, Örebro
  - Medicinklin, sekt för hematologi, Norrlands Universitetssjukhus, Umeå
  - Medicinklin, Akademiska sjukhuset, Uppsala

REFERENCES:
- [Derived] Mellqvist UH, Gimsing P, Hjertner O, Lenhoff S, Laane E, Remes K, Steingrimsdottir H, Abildgaard N, Ahlberg L, Blimark C, Dahl IM, Forsberg K, Gedde-Dahl T, Gregersen H, Gruber A, Guldbrandsen N, Haukas E, Carlson K, Kvam AK, Nahi H, Lindas R, Andersen NF, Turesson I, Waage A, Westin J; Nordic Myeloma Study Group. Bortezomib consolidation after autologous stem cell transplantation in multiple myeloma: a Nordic Myeloma Study Group randomized phase 3 trial. Blood. 2013 Jun 6;121(23):4647-54. doi: 10.1182/blood-2012-11-464503. Epub 2013 Apr 24. PMID 23616624